CLINICAL TRIAL: NCT05665309
Title: Interest of Pre-operative Use of 3D Printing for Endovascular Treatment of Unruptured Intracranial Aneurysms With Intrasaccular Flow Disruptor
Acronym: ILIAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/676
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With 3D anatomical model (Experimental): Surgery prepared using 3D anatomical model of the aneurysm
  Interventions: Procedure: 3D anatomical model of aneurysm
- Without 3D anatomical model (No Intervention): Surgery prepared without 3D anatomical model of the aneurysm (routine care)

INTERVENTIONS:
Procedure: 3D anatomical model of aneurysm — Surgery prepared with 3D anatomical model of aneurysm
  Arms: With 3D anatomical model

SUMMARY:
This is a preliminary randomised controlled trial comparing the use of pre-operative 3D models to select an intrasaccular flow disruptor for endovascular aneurysm cure.

DETAILED DESCRIPTION:
Patients will be randomised 3:1 either in the intervention or control group. Intervention consists of using the pre-operative Digital Subtraction Angiography (DSA) to create a 3D plastic model. This model is used to test different sizes of device. At the end of this pre-operative test a single device is recommended for the real procedure. The control group will use the current method for size selection (measurement of mean width and minimum height) on DSA.

ELIGIBILITY:
Inclusion Criteria:

* Intracranial aneurysm, suitable for a treatment by Woven Endobridge (WEB) device after multidisciplinary team decision
* Consent form signed
* The patient benefits from health insurance

Exclusion Criteria:

* Legal incapacity
* Women at risk of pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with successful procedure | Day 0
  Proportion of patients for which flow disruption succeeded at first intent, without any change of size required for WEB disruptor

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CHARBONNIER, MD, Principal Investigator — CHU de Besançon